CLINICAL TRIAL: NCT04937114
Title: Efficacy of Unidirectional Barbed Sutures on Various Outcomes in Mucogingival Procedures
Brief Title: Unidirectional Barbed Sutures in Mucogingival Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Primary Investigator, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/5/2020
Record Dates: First submitted 2021-06-17; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Wound Heal

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flap will be approximated using conventional, simple continuous suturing with barbed sutures (Experimental): After administration of adequate amount of local anesthesia, planned muco-gingival surgery will be performed and flap will be approximated using conventional, simple continuous suturing with unidirectional barbed sutures.
  Interventions: Procedure: Barbed suture
- Flap will be approximated using conventional, simple continuous suturing with conventional sutures (Active Comparator): After administration of adequate amount of local anesthesia, planned muco-gingival surgery will be performed and flap will be approximated using conventional, simple continuous suturing with conventional sutures.
  Interventions: Procedure: Barbed suture

INTERVENTIONS:
Procedure: Barbed suture — Experimental: Wound will be closed using unidirectional barbed sutures in muco-gingival surgeries Active Comparator: Wound will be closed using conventional sutures in muco-gingival surgeries

SUMMARY:
The aim of the study is to compare the efficacy of barbed suture with conventional suture in muco-gingival surgeries.

DETAILED DESCRIPTION:
Experimental: Main treatment group, flap will be approximated using conventional, simple continuous suturing with barbed sutures.

Comparator: In patients allocated to control group, flap will be approximated using conventional, simple continuous suturing with conventional sutures.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals within an age group of 20-50yrs with presence of attached gingiva, shallow vestibule and frenum interfering with the marginal gingiva.

Exclusion Criteria:

* Medically compromised patients.
* Subjects who underwent radiotherapy or chemotherapy in the past 12 months.
* Smokers

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
To assess primary wound closure | Baseline to 21days
  Primary wound closure and early wound healing by EHS at 7days,14days,21days

SECONDARY OUTCOMES:
To assess pain | Baseline to 21days
  Pain by Visual Analogous Scale immediately

CONTACTS AND LOCATIONS:
Locations (1):
- SVS Institute of Dental Sciences, Mahabubnagar, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No